CLINICAL TRIAL: NCT05945134
Title: Effects of Sit-to-stand Training With Interactive Feedback on Muscle Contraction Sequences and Weight Bearing Symmetry in Individuals With Chronic Stroke
Brief Title: Sit-to-stand Training With Interactive Feedback in Chronic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NYCU112081AE
Record Dates: First submitted 2023-07-03; First posted 2023-07-14 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-06

CONDITIONS: Stroke
Keywords: Interactive feedback; Muscle contraction sequence; Weight bearing symmetry; Sit-to-stand training; Chronic stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visual and auditory feedback STS training group (Experimental): The interactive interface of visual and auditory feedback system was designed using LabVIEW and integrated force plates for training. Signals from the pressure detectors of the seat and two force plates on the floor will be converted to the indication of the body weight distribution (indicated by the size of the two circles of both legs, larger circle represented the more weight beard on the leg) and the movement path of the overall center of pressure (indicated by a mobile solid dot).
  Interventions: Other: Visual and auditory feedback STS training
- Conventional STS training group (Active Comparator): Only verbal and visual cues which were commonly used by the therapist.
  Interventions: Other: Conventional STS training

INTERVENTIONS:
Other: Visual and auditory feedback STS training — 30 minutes per session, 3 sessions per week, for a total of 3 weeks. The visual and auditory feedback signals will be given throughout the sit-to-stand movement. As the size of circle representing the weight bearing gets more even, and the mobile dot indicating the overall center of pressure moves forward and approaches the midline, the auditory cues will get louder to indicate proximity to the target. It allows the participants to adjust and relearn the correct weight shifting and symmetry.
  The intensity will be adjusted based on different chair heights (e.g. 115%, 100%, 80% of lower leg length), various seat materials, and supported level of thigh (progressing from one-third of the length between the greater trochanter of the femur and the knee joint line to full support). The training program will be progressed according to the abilities of the participants.
  Arms: Visual and auditory feedback STS training group
Other: Conventional STS training — 30 minutes per session, 3 sessions per week, for a total of 3 weeks. All settings will be the same as the experimental group, except for the feedback. In the control group, the verbal cues will be given by the physical therapist and a mirror will be placed in front of the participant for visual feedback. During the sit-to-stand movement, participants will be asked to try to maintain the alignment in the midline.
  Arms: Conventional STS training group

SUMMARY:
The major problems of people with chronic stroke include muscle weakness, sensory alteration, and inter-muscular coordination impairment. Inter-muscular coordination impairment caused altered muscle contraction sequences and weight-bearing asymmetry during functional activities. Sit-to-stand (STS) training is often used to improve functional activities among post-stroke subjects. However, the improvement may come from compensatory movements. Using compensatory movement may cause muscle weakness in the affected side and increase fall risk. This study will develop a novel STS training system with interactive visual and audio feedback emphasizing weight transferring and weight bearing. The present study aims to investigate the effects of sit-to-stand training with interactive visual and audio feedback on muscle contraction sequences and weight bearing symmetry in individuals with chronic stroke.

DETAILED DESCRIPTION:
This is a prospective randomized single-blinded controlled trial with pre- and post-measurements. 20 individuals will be recruited, and randomly assigned to experimental or control group. Statistical data analysis will be done by SPSS 24.0. Baseline characteristics will be analyzed using independent t-test or Chi-square test. Repeated measures two-way analysis of variance (ANOVA) with Tukey's post-hoc analysis will be used for time-by-group comparisons. The significant level is set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke ≥ 6 months
* Mini-mental state examination (MMSE) ≥ 24 points
* Brunnstrom lower limb recovery stage: ≥ stage 3
* Be able to independently perform STS for at least 10 times
* Single STS >1.7 seconds
* Be able to walk ≥10 meters independently

Exclusion Criteria:

* Any other musculoskeletal, neurological and cardiovascular diseases
* Have visual or language impairments

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-15 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Sit to stand performance: change in onset time of muscle contraction sequences | 5 minutes, Change from baseline onset time at 3-week post-test
  Use the surface electromyography to evaluate the "onset" time (% MT, EMG activities ≥ 2 SD of the baseline for ≥100 ms) of different muscles recruited during sit to stand (rectus femoris, biceps femoris, gluteus maximus, tibialis anterior, gastrocnemius, and soleus)
Sit to stand performance: change in peak force time of muscle contraction sequences | 5 minutes, Change from baseline peak force time at 3-week post-test
  Use the surface electromyography to evaluate the "peak force" time (% MT, maximal EMG activities) of different muscles recruited during sit to stand (rectus femoris, biceps femoris, gluteus maximus, tibialis anterior, gastrocnemius, and soleus)
Sit to stand performance: change in offset time of muscle contraction sequences | 5 minutes, Change from baseline offset time at 3-week post-test
  Use the surface electromyography to evaluate the "offset" time (% MT, EMG activities < 2 SD of the baseline for ≥100 ms) of different muscles recruited during sit to stand (rectus femoris, biceps femoris, gluteus maximus, tibialis anterior, gastrocnemius, and soleus)
Sit to stand performance: change in weight bearing symmetry | 5 minutes, Change from baseline weight bearing symmetry at 3-week post-test
  Use the force plates to evaluate the "cumulative vertical force " (% of body weight), and calculate with the "asymmetry ratio" = |1-affected side/less affected side|
Sit to stand performance: change in COP sway pathway | 5 minutes, Change from baseline COP sway pathway at 3-week post-test
  Use the force plates to evaluate the total length (cm) of the moving pathway of the overall center of pressure in X or Y axis individually

SECONDARY OUTCOMES:
Sit to stand performance: change in sit to stand duration | 5 minutes, Change from baseline sit to stand duration at 3-week post-test
  Use the surface electromyography to evaluate the "movement time" (MT, sec), using the "offset time of the last activated muscle" - "onset time of the first activated muscle"
Gait performance: change in symmetry of gait speed | 5 minutes, Change from baseline symmetry of gait speed at 3-week post-test
  Use the GAITRite® system to evaluate gait speed (m/s) in comfortable speed (with/ without assisted device), and calculate with the "asymmetry ratio" = |1-affected side/less affected side|
Gait performance: change in symmetry of step length | 5 minutes, Change from baseline symmetry of step length at 3-week post-test
  Use the GAITRite® system to evaluate step length (m) in comfortable speed (with/ without assisted device), and calculate with the "asymmetry ratio" = |1-affected side/less affected side|
Gait performance: change in symmetry of step time | 5 minutes, Change from baseline symmetry of step time at 3-week post-test
  Use the GAITRite® system to evaluate step time (sec) in comfortable speed (with/ without assisted device), and calculate with the "asymmetry ratio" = |1-affected side/less affected side|

CONTACTS AND LOCATIONS:
Overall Officials: Ray-Yau Wang, PhD, Principal Investigator — rywang@nycu.edu.tw
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan